CLINICAL TRIAL: NCT04102150
Title: A Phase 2, Multicenter, Open-label, Single-arm Study of Valemetostat Tosylate (DS-3201b) in Patients With Relapsed or Refractory Adult T-cell Leukemia/Lymphoma
Brief Title: Valemetostat Tosylate (DS-3201b) Phase 2 Study in Relapsed or Refractory Adult T-cell Leukemia/Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS3201-A-J201; 194964 (Other: JAPIC CTI)
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Adult T-cell Leukemia/Lymphoma
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DS-3201b (Experimental)
  Interventions: Drug: Valemetostat Tosylate

INTERVENTIONS:
Drug: Valemetostat Tosylate — Once a day, 200 mg, oral administration
  Other Names: DS-3201b

SUMMARY:
This Phase 2 study will be conducted to assess the efficacy and safety of valemetostat tosylate (DS-3201b) in participants with relapsed or refractory adult T-cell leukemia/lymphoma (r/r ATL).

ELIGIBILITY:
Inclusion Criteria:

* Participants with relapsed or refractory adult T-cell leukemia/lymphoma (ATL) who have history of treatment with mogamulizumab or are mogamulizumab intolerant, contraindication after treatment with at least 1 medication regimen
* Aged ≥20 years or older at the time of signing the informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2
* At least 1 evaluable lesion
* Participants who have defined laboratory criteria
* Life expectancy ≥ 3 months

Exclusion Criteria:

* A presence of central nervous system involvement at the time of screening tests
* Have poorly controlled complication (eg. chronic congestive heart failure, unstable angina
* ≥ Grade 3 neuropathy
* QT interval corrected using Fridericia's method (QTcF) >470 ms
* Has an uncontrolled infection
* Participants who use corticosteroids over 10 mg/day
* Receipt of allogeneic hematopoietic stem cell transplantation
* History of, or concurrent, malignant tumors

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2021-04-24 (Actual); Study Completion 2024-10-27 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) assessed by central evaluation organization | Through the end of the study (within approximately 5 years)
  The percentage of participants who were assessed for best overall response, who achieved complete remission (CR), complete remission, unconfirmed (CRu) or partial remission (PR) by central evaluation organization.

SECONDARY OUTCOMES:
Overall response rate (ORR) assessed by investigator | Through the end of the study (within approximately 5 years)
  The percentage of participants who were assessed for best overall response, who achieved CR, CRu, or PR by investigator.
Best response per tumor lesions | Through the end of the study (within approximately 5 years)
  Best response in target lesions (nodal or extranodal lesions), peripheral blood lesions, and skin lesions.
Complete remission rate (CR rate) | Through the end of the study (within approximately 5 years)
  The percentage of participants who were assessed for best overall response, who achieved CR or CRu.
Tumor control rate (TCR) | Through the end of the study (within approximately 5 years)
  The percentage of participants who were assessed for best overall response, who achieved CR, CRu, PR or stable disease (SD).
Time to response (TTR) | Through the end of the study (within approximately 5 years)
  Period from the first day of DS-3201b dose to the first day of CR, CRu, or PR
Duration of response (DOR) | Through the end of the study (within approximately 5 years)
  Period from first CR, CRu, or PR to residual disease/progressive disease (RD/PD) or death.
Progression-free survival (PFS) | Through the end of the study (within approximately 5 years)
  Period from the first day of DS-3201b dose to the day of RD/PD or death.
Overall survival (OS) | Through the end of the study (within approximately 5 years)
  Period from the first day of DS-3201b dose to death.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (24):
- Japan (24):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Ehime University Hospital, Tōon-shi, Ehime
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Imamura General Hospital, Kagoshima, Kagoshima-ken
  - Kochi Medical School Hospital, Nankoku-shi, Kochi
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - National University Corporation Tohoku University Tohoku University Hospital, Sendai, Miyagi
  - University of Miyazaki Hospital, Miyazaki, Miyazaki
  - Local Incorporated Administrative Agency Sasebo City General Hospital, Sasebo-shi, Nagasaki
  - Okayama University Hospital, Okayama, Okayama-ken
  - University of the Ryukyus Hospital, Nakagami-gun, Okinawa
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Saga University Hospital, Saga, Saga-ken
  - Saitama Medical University International Medical Center, Hidaka-shi, Saitama
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - IMSUT Hospital, The Institute of Medical Science, The University of Tokyo, Minato-Ku, Tokyo
  - Kagoshima University Hospital, Kagoshima
  - Nagasaki University Hospital, Nagasaki

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: http://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Izutsu K, Makita S, Nosaka K, Yoshimitsu M, Utsunomiya A, Kusumoto S, Morishima S, Tsukasaki K, Kawamata T, Ono T, Rai S, Katsuya H, Ishikawa J, Yamada H, Kato K, Tachibana M, Kakurai Y, Adachi N, Tobinai K, Yonekura K, Ishitsuka K. An open-label, single-arm phase 2 trial of valemetostat for relapsed or refractory adult T-cell leukemia/lymphoma. Blood. 2023 Mar 9;141(10):1159-1168. doi: 10.1182/blood.2022016862. PMID 36150143